CLINICAL TRIAL: NCT05393895
Title: A Multi-Center, Double-Masked, Vehicle-Controlled, Evaluation of the Safety of CSF-1 in Presbyopic Subjects
Brief Title: An Evaluation of the Safety of CSF-1 in Presbyopic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orasis Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-150-0005
Record Dates: First submitted 2022-05-10; First posted 2022-05-26 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2022-12

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSF-1 (Experimental): One drop bilaterally twice daily for at least 6 weeks
  Interventions: Drug: CSF-1
- Vehicle (Placebo Comparator): One drop bilaterally twice daily for at least 6 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CSF-1 — One drop bilaterally twice daily for at least 6 weeks
  Other Names: Qlosi
  Arms: CSF-1
Drug: Vehicle — One drop bilaterally twice daily for at least 6 weeks
  Arms: Vehicle

SUMMARY:
This is a multi-center, double-masked, vehicle-controlled study. The purpose of the study is to evaluate the safety of CSF-1 compared with vehicle in presbyopic subjects. Subjects will be treated for at least 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have presbyopia

Exclusion Criteria:

* Have any contraindications to the study medications or diagnoses that would confound the study data

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Orasis Investigative Site, Newport Beach, California
  - Orasis Investigative Site, Petaluma, California
  - Orasis Investigative Site, Colorado Springs, Colorado
  - Orasis Investigative Site, Danbury, Connecticut
  - Orasis Investigative Site, Rock Island, Illinois
  - Orasis Investigative Site, Overland Park, Kansas
  - Orasis Investigative Site, Elizabeth City, North Carolina
  - Orasis Investigative Site, Fargo, North Dakota
  - Orasis Investigative Site, Cranberry Township, Pennsylvania
  - Orasis Investigative Site, Kingston, Pennsylvania
  - Orasis Investigative Site, Memphis, Tennessee
  - Orasis Investigative Site, Cedar Park, Texas

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | CSF-1 | Vehicle
Started | 118; 236 eyes | 60; 120 eyes
Completed | 110; 220 eyes | 50; 100 eyes
Not Completed | 8; 16 eyes | 10; 20 eyes
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | CSF-1 | Vehicle | Total
Number analyzed (Participants) | 118 | 60 | 178
Number analyzed (eyes) | 118 | 60 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (5.52) | 54.3 (5.55) | 54.3 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 44 | 115
  Male | 47 | 16 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 113 | 59 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 26 | 7 | 33
  White | 89 | 51 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 118 | 60 | 178
Iris Color [Count of Participants; unit: Participants]
  Light Iris Color | 63 | 33 | 96
  Dark Iris Color | 55 | 27 | 82
Manifest Refraction Spherical Equivalent (MRSE) [Number; unit: eyes] — MRSE: is the measure which allows to identify if a person is myopic (nearsighted) < -0.5D; emmetropic (normal refractive condition) between -0.5D to <= +0.75D: or hyperopic (farsighted) >+0.75D.
  For this measure, only 1 eye per participant was considered: the worst of both eyes or, if equal, the right eye.
  eyes
    -4.5D to <-0.5D | 24 | 14 | 38
    -0.5D to <= +0.75D | 67 | 35 | 102
    > +0.75D to +2.0D | 27 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events.
Description: As this is a safety study, no efficacy outcome has been defined.
Time Frame: Adverse events were collected over a period of at least 6 weeks and up to 21 weeks for the last participants exiting the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1 | Vehicle
Number analyzed (Participants) | 118 | 60
Participants | 43 | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of at least 6 weeks and up to 21 weeks for the last participants exiting the study.
Arm/Group | CSF-1 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/60
Other Adverse Events (participants affected / at risk) | 21/118 | 15/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CSF-1 (N=118) | Vehicle (N=60)
Conjunctival hyperaemia (Eye disorders) | 2 | 3 — All cases were mild in the CSF-1 and vehicle group.
Conjuctival papillae (Eye disorders) | 3 | 4 — All cases were mild in the CSF-1 and vehicle group.
Vision blurred (Eye disorders) | 5 | 5 — All cases were mild in the CSF-1 and vehicle group.
Instillation site pain (General disorders) | 21 | 0 — All cases were mild, with 80% of them being described as stinging or burning, lasting between a few seconds and a minute.
COVID-19 (Infections and infestations) | 1 | 3 — All cases were mild in the CSF-1 and vehicle group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05393895/Prot_SAP_000.pdf